CLINICAL TRIAL: NCT00113971
Title: A Randomized Phase II Pharmacokinetics/Pharmacodynamics Study of Epratuzumab in Patients With Systemic Lupus Erythematosus
Brief Title: Pharmacokinetics Study of Epratuzumab in Systemic Lupus Erythematosus (SLE)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SL0002 (IMMU-103-SLE-02)
Record Dates: First submitted 2005-06-10; First posted 2005-06-13 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: study of epratuzumab in systemic lupus erythematosus; systemic lupus erythematosus; SLE
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — epratuzumab

INTERVENTIONS:
Drug: epratuzumab

SUMMARY:
The goal of this study is to evaluate how epratuzumab is processed by the body (pharmacokinetics) and whether 2 dose levels of epratuzumab are safe and effective in patients with SLE.

DETAILED DESCRIPTION:
This study is planned to provide information on how the body processes epratuzumab and how epratuzumab affects the body when epratuzumab is given once weekly for 4 weeks in a row at one of 2 different dose levels. Additional information will be obtained related to the natural variability of disease activity in SLE patients.

ELIGIBILITY:
Inclusion Criteria:

* Has SLE by American College of Rheumatology revised criteria (meets >/= 4 criteria)
* Has had SLE for at least 6 months prior to study entry
* Has at least one elevated autoantibody level at study entry
* Has moderately active SLE disease at study entry in any body/organ system (Full criteria not present here due to length of considerations. The protocols should be consulted regarding the complete list of entry criteria.)

Exclusion criteria:

* Active Severe Lupus as defined by BILAG Index Level A in any body system or organ
* Allergy to human antibodies or Murine
* Prior therapy with other anti-B cell antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2005-04; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Evaluation of pharmacokinetic samples for epratuzumab levels and evaluation of adverse events, infusion reactions and other safety parameters.

SECONDARY OUTCOMES:
Evaluation of pharmacokinetic samples to assess immunogenicity and evaluation of post-treatment BILAG scores for initial efficacy and disease variability.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Barry, Study Director — UCB Pharma
Locations (3):
- United States (3):
  - Columbia Presbyterian Medical Center, New York, New York
  - Lupus Center of Excellence, Pittsburgh, Pennsylvania
  - Rheumatology Associates, Charleston, South Carolina

REFERENCES:
- [Background] Dorner T, Kaufmann J, Wegener WA, Teoh N, Goldenberg DM, Burmester GR. Initial clinical trial of epratuzumab (humanized anti-CD22 antibody) for immunotherapy of systemic lupus erythematosus. Arthritis Res Ther. 2006;8(3):R74. doi: 10.1186/ar1942. Epub 2006 Apr 21. PMID 16630358